CLINICAL TRIAL: NCT00628420
Title: A Randomized, Double Blind, Placebo Controlled, Single Oral Dose Study to Demonstrate the Safety, Tolerability, and Pharmacokinetics of ACP-104 (N-desmethylclozapine) in Schizophrenia, or Other Psychotic Disorders.
Brief Title: Safety Study of ACP-104: To Demonstrate the Safety, Tolerability, and Pharmacokinetics
Acronym: ACP-104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Stanley Medical Research Institute (Other); ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Carol A. Tamminga, MD, Professor, UT Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 082004-051
Record Dates: First submitted 2008-02-24; First posted 2008-03-05 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2008-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; N-desmethylclozapine; clozapine; psychosis; randomized; placebo studies
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Other): Patients recieved single low dose of ACP-104
  Interventions: Drug: ACP-104
- 2 (Other): Patients recieved a high dose of ACP-104
  Interventions: Drug: ACP-104
- 3 (Other): Patients recieved a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACP-104 — 25mg, 75mg, 125mg, 175mg, 225mg, or 275mg once a day for 2 weeks
  Arms: 1
Drug: ACP-104 — Patient will be given either 50mg, 100mg, 150mg, 200mg, 250mg, or 300mg daily for 2 weeks
  Arms: 2
Drug: Placebo — patients will be given a placebo: 25mg, 50mg, 75mg, 100mg, 125mg, 150mg, 175mg, 200mg, 225mg, 250mg, 275mg, or 300mg (to match the doses given) daily for 2 weeks.
  Other Names: cornstarch capsule
  Arms: 3

SUMMARY:
To determine the safety and tolerability of ACP-104 after oral administration of single doses in comparison with placebo to schizophrenia or other psychotic disorders.

DETAILED DESCRIPTION:
Thirty-six healthy patients with schizophrenia or psychotic disorders, each of whom will be drug-free at study initiation, will be admitted to the hospital and will each receive two doses of ACP-104, and one dose of placebo, orally every 3-5 days over a two-week period. The patients will be divided into six groups of up to six and minimum of 3 patients each. Group 1 will consist of six patients who will receive single 25mg and 50mg doses of ACP-104 and placebo in random, but rising dose, order over a two-week period. Data from group one will be collected to determine ACP-104's safety, tolerability, and pharmacokinetics. Group 2 will be enrolled in the study once study data from Group 1 has demonstrated the safety of ACP-104. Group 2 will receive a 25mg pre-conditioning dose of ACP-104. Following the pre-conditioning dose, 75mg and 100mg single doses of ACP-104 will be administered in random, but rising dose, order, over a two-week period. Group 3 will be enrolled in the study once study data from Group 2 has demonstrated the safety of ACP-104. Group 3 will receive a 25mg pre-conditioning dose of ACP-104. Following the pre-conditioning dose, 125mg and 150mg single doses of ACP-104 will be administered in random, but rising dose, order, over a two-week period. Group 4 will be enrolled in the study once study data from Group 3 has demonstrated the safety of ACP-104. Group 4 will receive a 25mg pre-conditioning dose of ACP-104. Following the pre-conditioning dose, 175mg and 200mg single doses of ACP-104 will be administered in random, but rising dose, order, over a two-week period. Group 5 will be enrolled in the study once study data from Group 4 has demonstrated the safety of ACP-104. Group 5 will receive a 25mg pre-conditioning dose of ACP-104. Following the pre-conditioning dose, 225mg and 250mg single doses of ACP-104 will be administered in random, but rising dose, order, over a two week period. Group 6 will be enrolled in the study once study data from Group 5 has demonstrated the safety of ACP-104. Group 6 will receive a 25mg pre-conditioning dose of ACP-104. Following the pre-conditioning dose, 275mg and 300mg single doses of ACP-104 will be administered in random, but rising dose, order, over a two-week period. Groups 1-6 will be monitored closely and safety procedures and evaluations will be performed on all medication days. Safety assessments will include: physical examinations, vital signs (3-positional blood pressure and pulse rate, respiration rate, and oral body temperature), clinical laboratory tests, ECGs (Electrocardiogram), coordination tests, questions about symptoms and side effects. Once all medication days have been completed, the condition of the patient will be assessed, and, at that time, it will be determined whether the patient's condition is suitable for release from the hospital or whether further monitoring of the patient's condition as an inpatient is needed.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, who have been surgically sterilized or at least 1 year post menopausal, in good health (based on medical history, physical examination, electrocardiograms, and clinical laboratory tests)
* Between 20 and 50 years old (inclusive)
* History of schizophrenia, schizoaffective disorder, bipolar with psychosis, major depression with psychosis, PTSD with psychosis, or psychosis NOS and not experiencing an acute exacerbation of severe psychosis
* Able to execute informed written consent
* Willing to follow dietary restrictions as outlined in Section 6.2 General and dietary restrictions,
* Willing to remain hospitalized for the in-patient portion of the study and return for follow up visit(s) as required by the protocol and as deemed necessary by principal investigator,
* Will be in need of treatment with an antipsychotic medication,
* Fluent and literate in English

Exclusion Criteria:

* Any patient that has received clozapine within the last three months, or any depot antipsychotic within the last six months,
* Likely allergy or insensitivity to ACP-104 or clozapine based on known allergies to drugs of the same class, or which in the opinion of the principle investigator, suggests an increased potential for an adverse hypersensitivity to ACP-104
* Any prior history of drug-induced leukopenia or neutropenia,
* Any prior history of neuroleptic malignant syndrome
* History of seizure, epilepsy, severe head injury, multiple sclerosis, or other known neurological condition
* Prior history of cardiovascular disease, including arrhythmia or myocarditis
* Abnormal pre-admission vital signs or clinical laboratory evaluations
* Any patient with a history, within the last three months, of alcohol and/or drug dependency or alcohol and/or drug abuse in the last month
* History of hepatic or renal disease
* Any patient scheduled to undergo any surgical procedure during the duration of the study,
* Any patient taking any concurrent medications for a major medical illness
* Any patient who has donated plasma or blood within 30 days before the first dose of study medication,
* Any patient who has received any known hepatic or renal clearance altering agents (e.g., erythromycin, cimetidine, barbiturates, phenothiazines, etc.) for a period of 3 months before the first dose of study medication
* Ingestion or use of any investigational medication or device within 3 months before the first dose of study medication
* Acute illness within 5 days before the first dose of study medication
* Mental capacity is limited to the extent that the patient cannot provide legal consent or understand information regarding the side effects or tolerance of the study drug
* Any patient judged by the principal investigator to be inappropriate for the study.

  * We do not have the resources necessary to properly study non-English speaking patients in this study. The need to provide such resources would be prohibitive to the successful completion of the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2005-01; Primary Completion 2006-11 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Veteran's Affairs Medical Center, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas